CLINICAL TRIAL: NCT01573624
Title: A Multi-center, Randomized, Double-blind, Dose-ranging Study to Evaluate GSK573719 in Combination With Fluticasone Furoate, Fluticasone Furoate Alone, and an Active Control of Fluticasone Furoate/Vilanterol Combination in Subjects With Asthma
Brief Title: Evaluate the Safety, Efficacy and Dose Response of GSK573719 in Combination With Fluticasone Furoate in Subjects With Asthma
Acronym: ILA115938
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Diagnostic
Other Study IDs: 115938
Record Dates: First submitted 2012-04-05; First posted 2012-04-09 (Estimated); Results first posted 2017-08-15 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-09

CONDITIONS: Asthma
Keywords: Fluticasone Furoate; Vilanterol; Adults; GSK573719; Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fluticasone Furoate (FF) (Active Comparator): 100mcg, inhaled
  Interventions: Drug: FF
- Fluticasone Furoate /Vilanterol (VI) (Active Comparator): 100/25mcg inhaled
  Interventions: Drug: FF/VI
- Fluticasone Furoate/GSK573719 (Experimental): 100/15.6-250mcg inhaled
  Interventions: Drug: FF/GSK573719

INTERVENTIONS:
Drug: FF/GSK573719 — 100/15.6
  Arms: Fluticasone Furoate/GSK573719
Drug: FF/GSK573719 — 100/31.25
  Arms: Fluticasone Furoate/GSK573719
Drug: FF/GSK573719 — 100/62.5
  Arms: Fluticasone Furoate/GSK573719
Drug: FF/GSK573719 — 100/125
  Arms: Fluticasone Furoate/GSK573719
Drug: FF/GSK573719 — 100/250
  Arms: Fluticasone Furoate/GSK573719
Drug: FF — 100
  Arms: Fluticasone Furoate (FF)
Drug: FF/VI — 100/25
  Arms: Fluticasone Furoate /Vilanterol (VI)

SUMMARY:
Brief Summary: The purpose of this study is to characterize the dose response of GSK573719 in combination with Fluticasone furoate 100mcg in patients with asthma. Treatment with inhaled Fluticasone furoate and Fluticasone furoate/Vilanterol are included as an active control.

Detailed Description: Long acting muscarinic receptor antagonists (anti-cholinergic bronhcodilator) exert their effects via distinct and complementary bronchodilator mechanisms on large and small airways. Most of the experience with older anti-cholinergics had been with acute use and little is known about their effect in chronic use in asthma. This is a multicenter, randomized, double-blind, crossover study to evaluate 5 doses of inhaled GSK573719 inhaled over 14 days in patients with asthma. Fluticasone furoate (100 mcg) and Fluticasone furoate/Vilanterol (100/59mcg) will be included as an active comparator. Each eligible subject will receive a sequence of 3 of 7 potential treatments for a total of 3 treatment periods per subject. The total duration of subject participation is approximately 14 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient
* 18 years of age or older at Visit 1
* Diagnosis of Asthma
* Male or eligible Female
* Pre-bronchodilator FEV1 of 40-80% of the predicted normal value at Visit 1
* Demonstrated reversibility by ≥12% and ≥200mL of FEV1 within 40 minutes following albuterol at Visit 1
* A need for regular controller therapy (i.e., inhaled corticosteroids alone or in combination with a long-acting beta-agonist, or leukotriene modifier etc.,) for a minimum of 8 weeks prior to Visit 1.

Exclusion Criteria:

* History of Life threatening asthma
* Respiratory infection not resolved
* Asthma exacerbation
* Concurrent respiratory disease
* Current Smokers
* Other diseases that are uncontrolled disease or disease state that, in the opinion of the investigator, would put the safety of the patient at risk through study participation or would confound the interpretation of the efficacy results if the condition/disease exacerbated during the study
* A positive Hepatitis B surface antigen or positive Hepatitis C antibody and/or HIV
* Visual clinical evidence of oropharyngeal candidiasis
* Drug or milk protein allergies
* Concomitant medications affecting course of asthma
* Use of any other investigational medication within 30 days or 5 drug half-lives (whichever is longer)
* Previous use of GSK573719
* Any disease preventing use of anticholinergics
* Any condition that impairs compliance with study protocol including visit schedule and completion of daily diaries
* Any subject with a history of alcohol or substance abuse
* Any affiliation with Investigator's site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2012-04-03 (Actual); Primary Completion 2013-02-04 (Actual); Study Completion 2013-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (23):
- United States (4):
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
- Argentina (3):
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, Mendoza
  - GSK Investigational Site, San Miguel de Tucumán
- Chile (5):
  - GSK Investigational Site, Valparaíso, Región de Valparaíso
  - GSK Investigational Site, Puente Alto - Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
  - GSK Investigational Site, Talca, Región Metro de Santiago
  - GSK Investigational Site, Santiago
- Russia (8):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Kazan'
  - GSK Investigational Site, Klin
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Ufa
  - GSK Investigational Site, Yaroslavl
- Thailand (3):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Khon Kaen
  - GSK Investigational Site, Nonthaburi

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Derived] Lee LA, Yang S, Kerwin E, Trivedi R, Edwards LD, Pascoe S. The effect of fluticasone furoate/umeclidinium in adult patients with asthma: a randomized, dose-ranging study. Respir Med. 2015 Jan;109(1):54-62. doi: 10.1016/j.rmed.2014.09.012. Epub 2014 Oct 2. PMID 25452139
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 115938 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 115938 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 115938 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 115938 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 115938 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 115938 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 115938 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted across 33 centres of 5 countries from 03 April 2012 to 04 February 2013 in adults aged 18 to 50 years with persistent asthma. Participants were randomized for 3 treatment periods of 2 weeks each.
Pre-assignment Details: A total of 706 participants were screened for this study designed in 3 period crossover, incomplete block manner; 523 participants entered 2-week open label run-in period where they received fluticasone furoate (FF) 100 micrograms (mcg) dry powder inhalation once daily. A total of 421 participants were randomized to double-blind treatment period.
Groups:
- FF 100 mcg First: Participants received a dose of FF 100 mcg via a dry powder inhaler (DPI) once daily in the morning for 14 days during the first treatment period of the 3 treatment periods as per their randomization sequence. The 3 treatment periods were separated by 2 washout periods of 12-14 days each. Participants were administered with open-label FF 100 mcg once daily in the morning via a DPI while on washout period. Participants were followed-up for 7 days post-treatment. Salbutamol metered-dose inhaler (MDI) was provided as the rescue medication.
- FF 100 mcg + UMEC 15.6 mcg First: Participants received fixed dose of FF 100 mcg and umeclidinium bromide (UMEC) 15.6 mcg via a DPI once daily in the morning for 14 days during the first treatment period of the 3 treatment periods as per their randomization sequence. The 3 treatment periods were separated by 2 washout periods of 12-14 days each. Participants were administered with open-label FF 100 mcg once daily in the morning via a DPI while on washout period. Participants were followed-up for 7 days post-treatment. Salbutamol MDI was provided as the rescue medication.
- FF 100 mcg + UMEC 31.25 mcg First: Participants received fixed dose of FF 100 mcg and UMEC 31.25 mcg via a DPI once daily in the morning for 14 days during the first treatment period of the 3 treatment periods as per their randomization sequence. The 3 treatment periods were separated by 2 washout periods of 12-14 days each. Participants were administered with open-label FF 100 mcg once daily in the morning via a DPI while on washout period. Participants were followed-up for 7 days post-treatment. Salbutamol MDI was provided as the rescue medication.
- FF 100 mcg + UMEC 62.5 mcg First: Participants received fixed dose of FF 100 mcg and UMEC 62.5 mcg via a DPI once daily in the morning for 14 days during the first treatment period of the 3 treatment periods as per their randomization sequence. The 3 treatment periods were separated by 2 washout periods of 12-14 days each. Participants were administered with open-label FF 100 mcg once daily in the morning via a DPI while on washout period. Participants were followed-up for 7 days post-treatment. Salbutamol MDI was provided as the rescue medication.
- FF 100 mcg + UMEC 125 mcg First: Participants received fixed dose of FF 100 mcg and UMEC 125 mcg via a DPI once daily in the morning for 14 days during the first treatment period of the 3 treatment periods as per their randomization sequence. The 3 treatment periods were separated by 2 washout periods of 12-14 days each. Participants were administered with open-label FF 100 mcg once daily in the morning via a DPI while on washout period. Participants were followed-up for 7 days post-treatment. Salbutamol MDI was provided as the rescue medication.
- FF 100 mcg + UMEC 250 mcg First: Participants received fixed dose of FF 100 mcg and UMEC 250 mcg via a DPI once daily in the morning for 14 days during the first treatment period of the 3 treatment periods as per their randomization sequence. The 3 treatment periods were separated by 2 washout periods of 12-14 days each. Participants were administered with open-label FF 100 mcg once daily in the morning via a DPI while on washout period. Participants were followed-up for 7 days post-treatment. Salbutamol MDI was provided as the rescue medication.
- FF 100 mcg + VI 25 mcg First: Participants received fixed dose of FF 100 mcg and vilanterol (VI) 25 mcg via a DPI once daily in the morning for 14 days during the first treatment period of the 3 treatment periods as per their randomization sequence. The 3 treatment periods were separated by 2 washout periods of 12-14 days each. Participants were administered with open-label FF 100 mcg once daily in the morning via a DPI while on washout period. Participants were followed-up for 7 days post-treatment. Salbutamol MDI was provided as the rescue medication.
Period: Period 1 : Treatment Period 1 (14 Days)
Arm/Group | FF 100 mcg First | FF 100 mcg + UMEC 15.6 mcg First | FF 100 mcg + UMEC 31.25 mcg First | FF 100 mcg + UMEC 62.5 mcg First | FF 100 mcg + UMEC 125 mcg First | FF 100 mcg + UMEC 250 mcg First | FF 100 mcg + VI 25 mcg First
Started | 64 | 62 | 60 | 63 | 58 | 55 | 59
Completed | 58 | 59 | 51 | 61 | 56 | 51 | 57
Not Completed | 6 | 3 | 9 | 2 | 2 | 4 | 2
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 4 | 3 | 6 | 1 | 2 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 0 | 0 | 2 | 0
Not completed — Protocol-defined stopping criteria | 0 | 0 | 1 | 1 | 0 | 1 | 1
Period: Period 2 : Washout Period 1 (12-14 Days)
Arm/Group | FF 100 mcg First | FF 100 mcg + UMEC 15.6 mcg First | FF 100 mcg + UMEC 31.25 mcg First | FF 100 mcg + UMEC 62.5 mcg First | FF 100 mcg + UMEC 125 mcg First | FF 100 mcg + UMEC 250 mcg First | FF 100 mcg + VI 25 mcg First
Started | 58 | 59 | 51 | 61 | 56 | 51 | 57
Completed | 57 | 58 | 48 | 56 | 56 | 48 | 55
Not Completed | 1 | 1 | 3 | 5 | 0 | 3 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 1 | 0 | 2 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 0 | 1
Not completed — Protocol-defined stopping criteria | 0 | 0 | 1 | 1 | 0 | 1 | 0
Period: Period 3 : Treatment Period 2 (14 Days)
Arm/Group | FF 100 mcg First | FF 100 mcg + UMEC 15.6 mcg First | FF 100 mcg + UMEC 31.25 mcg First | FF 100 mcg + UMEC 62.5 mcg First | FF 100 mcg + UMEC 125 mcg First | FF 100 mcg + UMEC 250 mcg First | FF 100 mcg + VI 25 mcg First
Started | 57 | 58 | 48 | 56 | 56 | 48 | 55
Completed | 50 | 52 | 45 | 55 | 53 | 43 | 55
Not Completed | 7 | 6 | 3 | 1 | 3 | 5 | 0
Not completed — Lack of Efficacy | 5 | 4 | 2 | 1 | 3 | 2 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 0 | 0 | 1 | 0
Not completed — Protocol-defined stopping criteria | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 4 : Washout Period 2 (12-14 Days)
Arm/Group | FF 100 mcg First | FF 100 mcg + UMEC 15.6 mcg First | FF 100 mcg + UMEC 31.25 mcg First | FF 100 mcg + UMEC 62.5 mcg First | FF 100 mcg + UMEC 125 mcg First | FF 100 mcg + UMEC 250 mcg First | FF 100 mcg + VI 25 mcg First
Started | 50 | 52 | 45 | 55 | 53 | 43 | 55
Completed | 49 | 48 | 43 | 53 | 52 | 41 | 52
Not Completed | 1 | 4 | 2 | 2 | 1 | 2 | 3
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 1 | 1 | 1 | 1 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Protocol-defined stopping criteria | 0 | 1 | 1 | 1 | 0 | 1 | 0
Period: Period 5 : Treatment Period 3 (14 Days)
Arm/Group | FF 100 mcg First | FF 100 mcg + UMEC 15.6 mcg First | FF 100 mcg + UMEC 31.25 mcg First | FF 100 mcg + UMEC 62.5 mcg First | FF 100 mcg + UMEC 125 mcg First | FF 100 mcg + UMEC 250 mcg First | FF 100 mcg + VI 25 mcg First
Started | 49 | 48 | 43 | 53 | 52 | 41 | 52
Completed | 46 | 47 | 43 | 53 | 51 | 39 | 48
Not Completed | 3 | 1 | 0 | 0 | 1 | 2 | 4
Not completed — Lack of Efficacy | 2 | 0 | 0 | 0 | 1 | 1 | 4
Not completed — Protocol Violation | 0 | 1 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 6 : Follow-up Period (7 Days)
Arm/Group | FF 100 mcg First | FF 100 mcg + UMEC 15.6 mcg First | FF 100 mcg + UMEC 31.25 mcg First | FF 100 mcg + UMEC 62.5 mcg First | FF 100 mcg + UMEC 125 mcg First | FF 100 mcg + UMEC 250 mcg First | FF 100 mcg + VI 25 mcg First
Started | 46 | 47 | 43 | 53 | 51 | 39 | 48
Completed | 45 | 47 | 43 | 53 | 49 | 38 | 48
Not Completed | 1 | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Treatments Combined: The participants received 3 of the 7 possible treatments during the 3 double blind treatment periods. Participants received study treatments in a crossover manner according to their randomization sequence. The 7 treatment regimens were, FF 100 mcg, FF 100 mcg + UMEC 15.6 mcg, FF 100 mcg + UMEC 31.25 mcg, FF 100 mcg + UMEC 62.5 mcg, FF 100 mcg + UMEC 125 mcg, FF 100 mcg + UMEC 250 mcg and FF 100 mcg + VI 25 mcg. The study treatments were administered via a DPI taken once daily in the morning for 14 days during each study period. The treatment periods were separated by 2 washout periods of 12-14 days each. During the two week run-in period and during the two washout period, participants were administered open-label FF 100 mcg once daily in the morning via a DPI. Participants were followed-up for 7 days post-treatment. Salbutamol MDI was provided as the rescue medication.
Arm/Group | All Treatments Combined
Number analyzed (Participants) | 421
Age, Continuous [Mean (Standard Deviation); unit: Years] | 47.5 (13.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 289
  Male | 132
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 36
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 367
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Model Predicted Change From Baseline Trough Force Expiratory Volume in 1 Second (FEV1)
Description: FEV1 is a lung function measure defined as the maximal amount of air that can be forcefully exhaled in one second. Highest FEV1 from the 3 acceptable spirometric efforts were recorded between 5.00 ante meridiem (AM) and 11.00 AM after withholding albuterol (salbutamol) at all visits for at least 4 hours. Baseline was defined as the pre- dose FEV1 value obtained on Day 1 and trough was defined as FEV1 value obtained 24 hours after morning dosing on Day 14 of each treatment period. Change from baseline value for each participant in each treatment period was the difference between the observed on-treatment value obtained 24 hours after morning dosing on Day 14 and the baseline value for that period. Slope-intercept on log dose model was used to predict trough FEV1 change from baseline for each of the FF+UMEC doses adjusted by FF 100 mcg alone. Mean value for the expected response and associated 95% confidence interval (CI) in change from baseline trough FEV1 is presented.
Time Frame: Baseline (Day 1) and Day 15 of each treatment period
Population: The primary endpoint was analyzed using Intent -to -Treat (ITT) Population defined as all participants randomized to treatment and who received at least one dose of study medication. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (95% Confidence Interval); unit: Litres (L)
Groups:
- FF 100 mcg + UMEC 15.6 mcg: Participants received fixed dose of FF 100 mcg and UMEC 15.6 mcg via a DPI once daily in the morning for 14 days in any one of the 3 treatment periods according to their randomization sequence. The 3 treatment periods were separated by 2 washout periods of 12-14 days each. Participants were administered with open-label FF 100 mcg once daily in the morning via a DPI while on washout period. Participants were followed-up for 7 days post-treatment. Salbutamol MDI was provided as the rescue medication.
- FF 100 mcg + UMEC 31.25 mcg: Participants received fixed dose of FF 100 mcg and UMEC 31.25 mcg via a DPI once daily in the morning for 14 days in any one of the 3 treatment periods according to their randomization sequence. The 3 treatment periods were separated by 2 washout periods of 12-14 days each. Participants were administered with open-label FF 100 mcg once daily in the morning via a DPI while on washout period. Participants were followed-up for 7 days post-treatment. Salbutamol MDI was provided as the rescue medication.
- FF 100 mcg + UMEC 62.5 mcg: Participants received fixed dose of FF 100 mcg and UMEC 62.5 mcg via a DPI once daily in the morning for 14 days in any one of the 3 treatment periods according to their randomization sequence. The 3 treatment periods were separated by 2 washout periods of 12-14 days each. Participants were administered with open-label FF 100 mcg once daily in the morning via a DPI while on washout period. Participants were followed-up for 7 days post-treatment. Salbutamol MDI was provided as the rescue medication.
- FF 100 mcg + UMEC 125 mcg: Participants received fixed dose of FF 100 mcg and UMEC 125 mcg via a DPI once daily in the morning for 14 days in any one of the 3 treatment periods according to their randomization sequence. The 3 treatment periods were separated by 2 washout periods of 12-14 days each. Participants were administered with open-label FF 100 mcg once daily in the morning via a DPI while on washout period. Participants were followed-up for 7 days post-treatment. Salbutamol MDI was provided as the rescue medication.
- FF 100 mcg + UMEC 250 mcg: Participants received fixed dose of FF 100 mcg and UMEC 250 mcg via a DPI once daily in the morning for 14 days in any one of the 3 treatment periods according to their randomization sequence. The 3 treatment periods were separated by 2 washout periods of 12-14 days each. Participants were administered with open-label FF 100 mcg once daily in the morning via a DPI while on washout period. Participants were followed-up for 7 days post-treatment. Salbutamol MDI was provided as the rescue medication.
Arm/Group | FF 100 mcg + UMEC 15.6 mcg | FF 100 mcg + UMEC 31.25 mcg | FF 100 mcg + UMEC 62.5 mcg | FF 100 mcg + UMEC 125 mcg | FF 100 mcg + UMEC 250 mcg
Number analyzed (Participants) | 154 | 146 | 150 | 155 | 150
Litres (L) | 0.0260 [-0.0098 to 0.0611] | 0.0320 [-0.0036 to 0.0679] | 0.0385 [-0.0011 to 0.0745] | 0.0444 [0.0067 to 0.0813] | 0.0510 [0.0139 to 0.0873]

2. Primary Outcome: Percentage of Chance That FF 100 mcg Alone Corrected Change From Baseline FEV1 Response Would Exceed a Target Response by Dose of UMEC Combined With FF 100 mcg
Description: FEV1 is a lung function measure defined as the maximal amount of air that can be forcefully exhaled in one second. Highest FEV1 from the 3 acceptable spirometric efforts were recorded between 5.00 AM and 11.00 AM after withholding albuterol (salbutamol) at all visits for at least 4 hours. Baseline was defined as the pre- dose FEV1 value obtained on Day 1 and trough was defined as FEV1 value obtained 24 hours after morning dosing on Day 14 of each treatment period. Change from baseline value for each participant in each treatment period was the difference between the observed on-treatment value obtained 24 hours after morning dosing on Day 14 and the baseline value for that period. Data is presented as percentage chance that FF 100 mcg alone corrected change from baseline trough FEV1 response would exceed a target response of 50 mL, 75 mL, 100 mL and 150 mL by doses of UMEC combined with FF 100 mcg.
Time Frame: Baseline (Day 1) and Day 15 of each treatment period
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Percentage chance
Arm/Group | FF 100 mcg + UMEC 15.6 mcg | FF 100 mcg + UMEC 31.25 mcg | FF 100 mcg + UMEC 62.5 mcg | FF 100 mcg + UMEC 125 mcg | FF 100 mcg + UMEC 250 mcg
Number analyzed (Participants) | 154 | 146 | 150 | 155 | 150
Percentage chance
  Target response of 50 mL | 9 | 17 | 27 | 37 | 52
  Target response of 75 mL | 0.5 | 1 | 2 | 5 | 10
  Target response of 100 mL | 0 | 0 | 0 | 0.2 | 0.2
  Target response of 150 mL | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Mean Change From Baseline in Trough FEV1 on Day 15 of Each of the 3 Treatment Periods
Description: FEV1 is a lung function measure defined as the maximal amount of air that can be forcefully exhaled in one second. The highest FEV1 from the 3 acceptable spirometric efforts were recorded between 5.00 AM and 11.00 AM after withholding albuterol (salbutamol) at all visits for at least 4 hours. Baseline was defined as the pre- dose FEV1 value obtained on Day 1 and trough was defined as the FEV1 value obtained 24 hours after morning dosing on Day 14 of each treatment period. The change from baseline value for each participant in each treatment period was the difference between the observed on-treatment value obtained 24 hours after morning dosing on Day 14 and the baseline value for that period. Analysis was done using a mixed model, including treatment, period, period baseline FEV1, and mean baseline FEV1 as fixed effects and participant as a random effect. A post hoc analysis was performed to confirm nullification of carry over effect of UMEC.
Time Frame: Baseline (Day 1) and Day 15 of each treatment period
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Litres (L)
Groups:
- FF 100 mcg: Participants received a dose of FF 100 mcg via a DPI once daily in the morning for 14 days in any one of the 3 treatment periods according to their randomization sequence. The 3 treatment periods were separated by 2 washout periods of 12-14 days each. Participants were administered with open-label FF 100 mcg once daily in the morning via a DPI while on washout period. Participants were followed-up for 7 days post-treatment. Salbutamol MDI was provided as the rescue medication.
- FF 100mcg + UMEC 15.6 mcg: Participants received fixed dose of FF 100 mcg and UMEC 15.6 mcg via a DPI once daily in the morning for 14 days in any one of the 3 treatment periods according to their randomization sequence. The 3 treatment periods were separated by 2 washout periods of 12-14 days each. Participants were administered with open-label FF 100 mcg once daily in the morning via a DPI while on washout period. Participants were followed-up for 7 days post-treatment. Salbutamol MDI was provided as the rescue medication.
- FF 100 mcg + VI 25 mcg: Participants received fixed dose of FF 100 mcg and VI 25 mcg via a DPI once daily in the morning for 14 days in any one of the 3 treatment periods according to their randomization sequence. The 3 treatment periods were separated by 2 washout periods of 12-14 days each. Participants were administered with open-label FF 100 mcg once daily in the morning via a DPI while on washout period. Participants were followed-up for 7 days post-treatment. Salbutamol MDI was provided as the rescue medication.
Arm/Group | FF 100 mcg | FF 100mcg + UMEC 15.6 mcg | FF 100 mcg + UMEC 31.25 mcg | FF 100 mcg + UMEC 62.5 mcg | FF 100 mcg + UMEC 125 mcg | FF 100 mcg + UMEC 250 mcg | FF 100 mcg + VI 25 mcg
Number analyzed (Participants) | 146 | 154 | 146 | 150 | 155 | 150 | 147
Litres (L) | 0.120 (0.0175) | 0.145 (0.0170) | 0.152 (0.0174) | 0.145 (0.0172) | 0.174 (0.0170) | 0.175 (0.0172) | 0.198 (0.0174)
Statistical Analysis 1: Comparison: FF 100 mcg vs FF 100mcg + UMEC 15.6 mcg; No pairwise comparisons between doses of FF + UMEC and FF alone were done unless overall F-test for treatment effect was statistically significant at 5% level. Multiplicity across these comparisons was controlled using a step-down closed testing procedure, whereby statistical comparison of the highest dose of FF + UMEC and FF alone was initially performed, and subsequent comparisons at lower doses continued in a step-down manner if preceding comparison was statistically significant at 5% level; Test type: Superiority or Other; p = 0.264, Mixed Models Analysis; Mean Difference (Net) = 0.026, 95% CI 2-sided [-0.019 to 0.071]
Statistical Analysis 2: Comparison: FF 100 mcg vs FF 100 mcg + UMEC 31.25 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.165, Mixed Models Analysis; Mean Difference (Net) = 0.033, 95% CI 2-sided [-0.013 to 0.079]
Statistical Analysis 3: Comparison: FF 100 mcg vs FF 100 mcg + UMEC 62.5 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.271, Mixed Models Analysis; Mean Difference (Net) = 0.026, 95% CI 2-sided [-0.020 to 0.071]
Statistical Analysis 4: Comparison: FF 100 mcg vs FF 100 mcg + UMEC 125 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.018, Mixed Models Analysis; Mean Difference (Net) = 0.055, 95% CI 2-sided [0.010 to 0.100]
Statistical Analysis 5: Comparison: FF 100 mcg vs FF 100 mcg + UMEC 250 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.018, Mixed Models Analysis; Mean Difference (Net) = 0.055, 95% CI 2-sided [0.010 to 0.101]
Statistical Analysis 6: Comparison: FF 100 mcg vs FF 100 mcg + VI 25 mcg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.078, 95% CI 2-sided [0.032 to 0.124]
Statistical Analysis 7: Comparison: FF 100mcg + UMEC 15.6 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p = 0.023, Mixed Models Analysis; Mean Difference (Net) = -0.052, 95% CI 2-sided [-0.097 to -0.007]
Statistical Analysis 8: Comparison: FF 100 mcg + UMEC 31.25 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p = 0.051, Mixed Models Analysis; Mean Difference (Net) = -0.045, 95% CI 2-sided [-0.091 to 0.000]
Statistical Analysis 9: Comparison: FF 100 mcg + UMEC 62.5 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p = 0.023, Mixed Models Analysis; Mean Difference (Net) = -0.053, 95% CI 2-sided [-0.098 to -0.007]
Statistical Analysis 10: Comparison: FF 100 mcg + UMEC 125 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p = 0.306, Mixed Models Analysis; Mean Difference (Final Values) = -0.023, 95% CI 2-sided [-0.068 to 0.021]
Statistical Analysis 11: Comparison: FF 100 mcg + UMEC 250 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p = 0.330, Mixed Models Analysis; Mean Difference (Net) = -0.023, 95% CI 2-sided [-0.068 to 0.023]

4. Secondary Outcome: Mean Change From Baseline in Daily Morning (Pre-dose and Pre-rescue Bronchodilator) Peak Expiratory Flow (PEF) of Each Treatment Period
Description: PEF is a measure of lung function and measures how fast a person can breathe out. Morning PEF was measured pre-dose and pre- rescue bronchodilator use with an electronic Peak Flow Meter. Participants were issued an electronic diary (eDiary) for daily use throughout the study and instructed on how to complete it. Best of 3 attempts were recorded in eDiary. Mean change from baseline was calculated where, baseline was defined as the measurement from (Week 0), includes Day 1 and six days immediately preceding Day 1 for each treatment period. The change from baseline values for each participant in each treatment period were differences between on-treatment week (last 7 days of each treatment period) values and baseline week. Analysis was done using a mixed model, including treatment, period, period baseline morning PEF and mean baseline morning PEF as fixed effects and participant as a random effect. A post hoc analysis was performed to confirm nullification of carry over effect of UMEC.
Time Frame: Baseline (Week 0) and last 7 days of each treatment period
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Litres per min (L/min)
Arm/Group | FF 100 mcg | FF 100 mcg + UMEC 15.6 mcg | FF 100 mcg + UMEC 31.25 mcg | FF 100 mcg + UMEC 62.5 mcg | FF 100 mcg + UMEC 125 mcg | FF 100 mcg + UMEC 250 mcg | FF 100 mcg + VI 25 mcg
Number analyzed (Participants) | 159 | 159 | 156 | 155 | 158 | 159 | 156
Litres per min (L/min) | -2.9 (2.44) | 13.0 (2.44) | 14.5 (2.46) | 15.7 (2.47) | 20.0 (2.44) | 19.0 (2.44) | 24.1 (2.46)
Statistical Analysis 1: Comparison: FF 100 mcg vs FF 100 mcg + UMEC 15.6 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 15.9, 95% CI 2-sided [9.5 to 22.3]
Statistical Analysis 2: Comparison: FF 100 mcg vs FF 100 mcg + UMEC 31.25 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 17.4, 95% CI 2-sided [10.9 to 23.9]
Statistical Analysis 3: Comparison: FF 100 mcg vs FF 100 mcg + UMEC 62.5 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 18.6, 95% CI 2-sided [12.1 to 25.1]
Statistical Analysis 4: Comparison: FF 100 mcg vs FF 100 mcg + UMEC 125 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 22.9, 95% CI 2-sided [16.5 to 29.4]
Statistical Analysis 5: Comparison: FF 100 mcg vs FF 100 mcg + UMEC 250 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 22.0, 95% CI 2-sided [15.5 to 28.4]
Statistical Analysis 6: Comparison: FF 100 mcg vs FF 100 mcg + VI 25 mcg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 27.0, 95% CI 2-sided [20.6 to 33.5]
Statistical Analysis 7: Comparison: FF 100 mcg + UMEC 15.6 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -11.2, 95% CI 2-sided [-17.6 to -4.7]
Statistical Analysis 8: Comparison: FF 100 mcg + UMEC 31.25 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis; Mean Difference (Net) = -9.6, 95% CI 2-sided [-16.1 to -3.1]
Statistical Analysis 9: Comparison: FF 100 mcg + UMEC 62.5 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p = 0.012, Mixed Models Analysis; Mean Difference (Net) = -8.4, 95% CI 2-sided [-14.9 to -1.9]
Statistical Analysis 10: Comparison: FF 100 mcg + UMEC 125 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p = 0.209, Mixed Models Analysis; Mean Difference (Net) = -4.1, 95% CI 2-sided [-10.6 to 2.3]
Statistical Analysis 11: Comparison: FF 100 mcg + UMEC 250 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p = 0.124, Mixed Models Analysis; Mean Difference (Net) = -5.1, 95% CI 2-sided [-11.6 to 1.4]

5. Secondary Outcome: Mean Change From Baseline in Daily Evening (Pre-dose and Pre-rescue Bronchodilator) PEF of Each Treatment Period
Description: PEF is a measure of lung function and measures how fast a person can breathe out. Evening PEF was measured pre-dose and pre-rescue bronchodilator use with an electronic Peak Flow Meter. Participants were issued an electronic diary (eDiary) for daily use throughout the study and instructed on how to complete it. Best of 3 attempts were recorded in eDiary. Mean change from baseline was calculated where, baseline was defined as the measurement from (Week 0), includes Day 1 and seven days immediately preceding Day 1 for each treatment period. The change from baseline values for each participant in each treatment period were differences between on-treatment week (last 7 days of each treatment period) values and baseline week. Analysis was done using a mixed model, including treatment, period, period baseline evening PEF and mean baseline evening PEF as fixed effects and participant as a random effect. A post hoc analysis was performed to confirm nullification of carry over effect of UMEC.
Time Frame: Baseline (Week 0) and last 7 days of each treatment period
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | FF 100 mcg | FF 100 mcg + UMEC 15.6 mcg | FF 100 mcg + UMEC 31.25 mcg | FF 100 mcg + UMEC 62.5 mcg | FF 100 mcg + UMEC 125 mcg | FF 100 mcg + UMEC 250 mcg | FF 100 mcg + VI 25 mcg
Number analyzed (Participants) | 160 | 157 | 156 | 154 | 157 | 157 | 153
L/min | -5.2 (2.51) | 11.1 (2.53) | 12.1 (2.54) | 16.0 (2.56) | 23.7 (2.52) | 17.7 (2.52) | 21.4 (2.58)
Statistical Analysis 1: Comparison: FF 100 mcg vs FF 100 mcg + UMEC 15.6 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 16.2, 95% CI 2-sided [9.5 to 22.9]
Statistical Analysis 2: Comparison: FF 100 mcg vs FF 100 mcg + UMEC 31.25 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 17.2, 95% CI 2-sided [10.5 to 24.0]
Statistical Analysis 3: Comparison: FF 100 mcg vs FF 100 mcg + UMEC 62.5 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 21.2, 95% CI 2-sided [14.4 to 28.0]
Statistical Analysis 4: Comparison: FF 100 mcg vs FF 100 mcg + UMEC 125 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 28.8, 95% CI 2-sided [22.1 to 35.5]
Statistical Analysis 5: Comparison: FF 100 mcg vs FF 100 mcg + UMEC 250 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 22.9, 95% CI 2-sided [16.2 to 29.6]
Statistical Analysis 6: Comparison: FF 100 mcg vs FF 100 mcg + VI 25 mcg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 26.6, 95% CI 2-sided [19.8 to 33.4]
Statistical Analysis 7: Comparison: FF 100 mcg + UMEC 15.6 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p = 0.003, Mixed Models Analysis; Mean Difference (Net) = -10.3, 95% CI 2-sided [-17.2 to -3.5]
Statistical Analysis 8: Comparison: FF 100 mcg + UMEC 31.25 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p = 0.007, Mixed Models Analysis; Mean Difference (Net) = -9.3, 95% CI 2-sided [-16.2 to -2.5]
Statistical Analysis 9: Comparison: FF 100 mcg + UMEC 62.5 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p = 0.126, Mixed Models Analysis; Mean Difference (Net) = -5.4, 95% CI 2-sided [-12.3 to 1.5]
Statistical Analysis 10: Comparison: FF 100 mcg + UMEC 125 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p = 0.523, Mixed Models Analysis; Mean Difference (Net) = 2.2, 95% CI [-4.6 to 9.1]
Statistical Analysis 11: Comparison: FF 100 mcg + UMEC 250 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p = 0.290, Mixed Models Analysis; Mean Difference (Net) = -3.7, 95% CI 2-sided [-10.5 to 3.1]

6. Secondary Outcome: Mean Change From Baseline in Rescue Albuterol/Salbutamol Use of Each Treatment Period.
Description: Short-Acting Beta2-Agonists albuterol/salbutamol was provided to participants as rescue medication, to use in morning and evening. Participants recorded number of puffs of salbutamol MDI used in last 24 hours (sum of night time and day time puffs) daily for relief of symptoms in eDiary. Mean change from baseline was calculated where, baseline was defined as measurement from (Week 0), includes Day 1 and six days immediately preceding Day 1 (for night time puffs) and seven days (for day time puffs) for each treatment period. Change from baseline values for each participant in each treatment period were differences between on-treatment week (last 7 days of each treatment period) values and the baseline week. Analysis was done using a mixed model, including treatment, period, period baseline rescue albuterol use, and mean baseline rescue albuterol use as fixed effects and participant as random effect. A post hoc analysis was performed to confirm nullification of carry over effect of UMEC.
Time Frame: Baseline (Week 0) and last 7 days of each treatment period
Population: ITT Population. Only those participants with data available at the indicated time points were analyzed.
Measure: Least Squares Mean (Standard Error); unit: Number of puffs
Arm/Group | FF 100 mcg | FF 100 mcg + UMEC 15.6 mcg | FF 100 mcg + UMEC 31.25 mcg | FF 100 mcg + UMEC 62.5 mcg | FF 100 mcg + UMEC 125 mcg | FF 100 mcg + UMEC 250 mcg | FF 100 mcg + VI 25 mcg
Number analyzed (Participants) | 158 | 151 | 152 | 151 | 153 | 157 | 151
Number of puffs | -0.2 (0.09) | -0.4 (0.09) | -0.4 (0.09) | -0.3 (0.09) | -0.5 (0.09) | -0.4 (0.09) | -0.6 (0.09)
Statistical Analysis 1: Comparison: FF 100 mcg vs FF 100 mcg + UMEC 15.6 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.036, Mixed Models Analysis; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.5 to 0.0]
Statistical Analysis 2: Comparison: FF 100 mcg vs FF 100 mcg + UMEC 31.25 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.064, Mixed Models Analysis; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.5 to 0.0]
Statistical Analysis 3: Comparison: FF 100 mcg vs FF 100 mcg + UMEC 62.5 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.335, Mixed Models Analysis; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.3 to 0.1]
Statistical Analysis 4: Comparison: FF 100 mcg vs FF 100 mcg + UMEC 125 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.012, Mixed Models Analysis; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to -0.1]
Statistical Analysis 5: Comparison: FF 100 mcg vs FF 100 mcg + UMEC 250 mcg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.023, Mixed Models Analysis; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.5 to 0.0]
Statistical Analysis 6: Comparison: FF 100 mcg vs FF 100 mcg + VI 25 mcg; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.4, 95% CI 2-sided [-0.7 to -0.2]
Statistical Analysis 7: Comparison: FF 100 mcg + UMEC 15.6 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p = 0.104, Mixed Models Analysis; Mean Difference (Net) = 0.2, 95% CI 2-sided [0.0 to 0.4]
Statistical Analysis 8: Comparison: FF 100 mcg + UMEC 31.25 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p = 0.062, Mixed Models Analysis; Mean Difference (Net) = 0.2, 95% CI 2-sided [0.0 to 0.5]
Statistical Analysis 9: Comparison: FF 100 mcg + UMEC 62.5 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p = 0.006, Mixed Models Analysis; Mean Difference (Net) = 0.3, 95% CI 2-sided [0.1 to 0.6]
Statistical Analysis 10: Comparison: FF 100 mcg + UMEC 125 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p = 0.217, Mixed Models Analysis; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.1 to 0.4]
Statistical Analysis 11: Comparison: FF 100 mcg + UMEC 250 mcg vs FF 100 mcg + VI 25 mcg; No adjustments were made for comparisons between doses of FF + UMEC and FF + VI; Test type: Superiority or Other; p = 0.143, Mixed Models Analysis; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.1 to 0.4]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from the start of study treatment (Visit 3) up to the follow-up (Visit 12, held 7 days from the Day 15 of treatment period 3 [Visit 11]). AE's and SAE's were reported for the treatment period only ( Visit 11 [up to Day 15 of the treatment period 3]).
Description: ITT Population was used.
Arm/Group | FF 100 mcg | FF 100 mcg + UMEC 15.6 mcg | FF 100 mcg + UMEC 31.25 mcg | FF 100 mcg + UMEC 62.5 mcg | FF 100 mcg + UMEC 125 mcg | FF 100 mcg + UMEC 250 mcg | FF 100 mcg + VI 25 mcg
All-Cause Mortality (participants affected / at risk) | 0/187 | 0/183 | 0/179 | 0/180 | 0/176 | 0/186 | 0/172
Serious Adverse Events (participants affected / at risk) | 0/187 | 0/183 | 1/179 | 0/180 | 0/176 | 0/186 | 1/172
Other Adverse Events (participants affected / at risk) | 3/187 | 4/183 | 2/179 | 5/180 | 4/176 | 7/186 | 6/172
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FF 100 mcg (N=187) | FF 100 mcg + UMEC 15.6 mcg (N=183) | FF 100 mcg + UMEC 31.25 mcg (N=179) | FF 100 mcg + UMEC 62.5 mcg (N=180) | FF 100 mcg + UMEC 125 mcg (N=176) | FF 100 mcg + UMEC 250 mcg (N=186) | FF 100 mcg + VI 25 mcg (N=172)
Cholecystitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FF 100 mcg (N=187) | FF 100 mcg + UMEC 15.6 mcg (N=183) | FF 100 mcg + UMEC 31.25 mcg (N=179) | FF 100 mcg + UMEC 62.5 mcg (N=180) | FF 100 mcg + UMEC 125 mcg (N=176) | FF 100 mcg + UMEC 250 mcg (N=186) | FF 100 mcg + VI 25 mcg (N=172)
Headache (Nervous system disorders) | 3 | 4 | 2 | 5 | 4 | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.